CLINICAL TRIAL: NCT04011813
Title: Official Title: Hypotaurine Supplementation in Freezing and Preparation Media Improves Human Sperm DeoxyriboNucleic Acid (DNA) and Fertilizing Ability
Brief Title: Hypotaurine Supplementation Benefits in Cryopreservation
Acronym: HYPOTAURINE
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Université d'Auvergne, Institut National de la Santéet de la Recherche Médicale (Unknown); Université d'Auvergne, Centre National de la Recherche Scientifique (Unknown); University Hospital, Clermont-Ferrand, Hematology laboratory (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2014 HYPOTAURINE
Record Dates: First submitted 2019-06-21; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Cryopreservation; Human Spermatozoa Parameters; Hypotaurine Supplementation; Spermatozoa DNA Alterations
Keywords: cryopreservation; density gradient centrifugation; DNA fragmentation, oxidation, chromatin packaging; antioxidant hypotaurine supplementation; cryo-capacitation; human spermatozoa fertilizing ability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control arm, "H-": semen treated without hypotaurine supplementation in density gradient centrifugation, washing and cryopreservation media
- Experimental arm, "H+": semen treated with a 50mM hypotaurine supplementation in density gradient centrifugation, washing and cryopreservation media
  Interventions: Other: Hypotaurine : antioxidant and osmoregulator

INTERVENTIONS:
Other: Hypotaurine : antioxidant and osmoregulator — Hypotaurine has protective effects on sperm motility, capacitation and acrosome reaction and reduces apoptotic markers.
  Hypotaurine (50mM) was added in density gradient centrifugation, washing and cryopreservation media washing and cryopreservation media before spermatozoa freezing
  Groups: Experimental arm, "H+"

SUMMARY:
Although it is widely used, slow freezing can induce strong functional and nuclear spermatic alterations reducing the chances of pregnancy. The study objective is to determinate the effects of the combination of hypotaurine supplementation and spermatozoa selection by Density Gradient Centrifugation (DGC) on human sperm functions and DNA quality during a freezing-thawing cycle.

DETAILED DESCRIPTION:
This prospective study was performed on surplus semen after a density gradient centrifugation-frozen-thawing cycle. Samples were obtained from men undergoing routine semen analysis at the Center for Reproductive Medicine. Spermatozoa were selected by density gradient centrifugation, washed and frozen using a programmable device. Each step was performed in parallel with (H+ arm) or without (H- arm) 50mM hypotaurine supplementation. After thawing, investigator team compared for both conditions the total and progressive mobility, vitality, integrity of the acrosome, markers of Protein Kinase A (PKA) dependent capacitation intracellular signaling pathway and nuclear quality by measuring chromatin packaging, DNA fragmentation and oxidation and vacuoles presence in the spermatozoa head.

ELIGIBILITY:
Inclusion Criteria:

* None

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men undergoing routine semen analysis at the Center for Reproductive Medicine
Enrollment: 33 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
chromatin packaging labelled using aniline blue and chromomycin A3 | Day 0
  Comparison after a cycle of freezing-thawing for both conditions, with or without hypotaurine supplementation of chromatin packaging labelled using aniline blue and chromomycin A3
DNA fragmentation using TUNEL assay | Day 0
  Comparison after a cycle of freezing-thawing for both conditions, with or without hypotaurine supplementation of DNA fragmentation using TUNEL assay
DNA oxidation assessed by 8-OHdG immunodetections | Day 0
  Comparison after a cycle of freezing-thawing for both conditions, with or without hypotaurine supplementation of DNA oxidation assessed by 8-OHdG immunodetections
vacuoles presence in the spermatozoa head using Motile Sperm Organelle Morphology Examination (MSOME) | Day 0
  Comparison after a cycle of freezing-thawing for both conditions, with or without hypotaurine supplementation of vacuoles presence in the spermatozoa head using Motile Sperm Organelle Morphology Examination (MSOME)

SECONDARY OUTCOMES:
vitality using Eosin Nigrosin | Day 0
  Comparison after a cycle of freezing-thawing for both conditions, with or without hypotaurine supplementation of vitality using Eosin Nigrosin
motility total and progressive | Day 0
  Comparison after a cycle of freezing-thawing for both conditions, with or without hypotaurine supplementation of motility total and progressive
integrity of the acrosome using Fluorescein IsoThioCyanate-Pisum Sativum Agglutinin (FITC-PSA) labelling | Day 0
  Comparison after a cycle of freezing-thawing for both conditions, with or without hypotaurine supplementation of integrity of the acrosome using Fluorescein IsoThioCyanate-Pisum Sativum Agglutinin (FITC-PSA) labelling
markers of PKA-dependent capacitation intracellular signaling pathway assessing western blot | Day 0
  Comparison after a cycle of freezing-thawing for both conditions, with or without hypotaurine supplementation of markers of PKA-dependent capacitation intracellular signaling pathway assessing western blot

CONTACTS AND LOCATIONS:
Overall Officials: Florence BRUGNON, MD, PhD, Principal Investigator — University Hospital, Clermont-Ferrand

REFERENCES:
- [Derived] Pons-Rejraji H, Vorilhon S, Difrane A, Dollet S, Bourgne C, Berger M, Chaput L, Pereira B, Bouche C, Drevet JR, Brugnon F. Beneficial effects of hypotaurine supplementation in preparation and freezing media on human sperm cryo-capacitation and DNA quality. Basic Clin Androl. 2021 Nov 4;31(1):26. doi: 10.1186/s12610-021-00144-6. PMID 34732137